CLINICAL TRIAL: NCT06977126
Title: First-in Human Clinical Trial Assessing Porphysome Nanoparticles for Biodistribution and Safety, in Imaging of Advanced Metastatic Gynaecological Cancers
Brief Title: Study to Assess the Safety and Effects of Porphysome Nanoparticles for Imaging in Gynaecological Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OZUHN-005
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gynecological Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PORPHYSOMES and 64Cu-PORPHYSOMES (64Cu-PS) (Experimental): Participants will receive one dose of 64Cu-PS with one dose of unlabelled PS (except for cohort 1) by intravenous (IV) route on Day 1.
  Interventions: Drug: PORPHYSOMES; Drug: 64Cu-PORPHYSOMES

INTERVENTIONS:
Drug: PORPHYSOMES — Pegylated porphyrin-lipid conjugate-containing nanoparticle suspension
Drug: 64Cu-PORPHYSOMES — Pegylated Copper-64 labelled porphyrin-lipid conjugate-containing nanoparticle suspension

SUMMARY:
This is an open-label, first-in-human, dose escalation study evaluating investigational drug PORPHYSOSMES (PS, pegylated porphyrin-lipid conjugate-containing nanoparticle suspension) and 64Cu-PORPHYSOMES (64Cu-PS, pegylated Copper-64 labelled porphyrin-lipid conjugate-containing nanoparticle suspension) for PET/CT imaging assessments in patients with metastatic/advanced gynecological tumors.

ELIGIBILITY:
Inclusion Criteria:

* Female patients age ≥ 18 years.
* Life expectancy of >3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Histologically confirmed metastatic advanced gynecological cancer. All epithelial subtypes are permitted. Patients receiving standard of care oncological treatment (i.e. chemotherapy and/or radiation) will be included.
* Patient is able to understand and is willing to sign a written informed consent document prior to registration/enrollment on to study.
* Patient is willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Patients of childbearing potential (as assessed by their local Investigator) and their partners who are sexually active must agree to the use of 2 highly effective forms of contraception throughout the period of study treatment and for 12 months after last dose of study drug.
* Baseline corrected QT (QTc) interval prolongation < 470 milliseconds.
* Within 8 days of the proposed enrollment patients must have adequate organ function.

Exclusion Criteria:

* Patient is a candidate for therapy with curative intent.
* Patient has a contraindication to PET/CT imaging, including, but not limited to, phobias associated with imaging (e.g. claustrophobia) and those who cannot lie still in the supine position for at least 20 minutes.
* Patients receiving nuclear medicine scans with other radiopharmaceutical agents (ex: 18F-FDG or other) during the study's exclusionary period will be excluded from the study.
* Patients with known myelodysplastic syndrome/acute myeloid leukemia.
* Treatment with an investigational drug within 15 days prior to study registration.
* Patients must not receive any other oncological treatments, including chemotherapy and/or radiation, within 2 weeks before starting study drug administration (and for 28 days after study drug administration).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
* Patients with a known active COVID-19 infection at the time of registration/enrollment.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the subject inappropriate for entry into this study.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection requiring IV antibiotics, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast-feeding women.
* Unresolved toxicity > CTCAE grade 1 from previous anti-cancer therapies, including radiotherapy, with exception.
* Retinopathy ≥ grade 2.
* Patients with porphyria.
* Patients that have undergone a splenectomy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2027-11-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | 1 year
  To determine the recommended dose of PORPHYSOME.

SECONDARY OUTCOMES:
Incidence of AEs | 1 year
  To evaluate the safety and tolerability of PS administration in subjects with advanced metastatic gynaecological cancers.
Tissue distribution and tumour uptake kinetics | 1 year
  To identify the tissue distribution and tumour uptake of escalating PS drug doses.
Concentration-time curves | 1 year
  To identify the plasma pharmacokinetic profiles of escalating PS drug doses.
Image- and model-based organ dosimetry | 1 year
  To estimate the radiation dosimetry of 64Cu-PS in healthy organ structures.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, MD, Principal Investigator — Princess Margaret Cancer Centre/University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No